CLINICAL TRIAL: NCT05515536
Title: Long-Term Open-Label Study to Assess the Safety and Efficacy of Vatiquinone in Patients With Friedreich Ataxia
Brief Title: A Study to Assess the Safety and Efficacy of Vatiquinone in Participants With Friedreich Ataxia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC743-NEU-003e-FA; 2022-002668-65 (EudraCT Number); 2024-516505-23-00 (Other: EU CT Number)
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vatiquinone (Experimental): Participants with FA who were previously treated with vatiquinone at an investigational site and completed participation in a prior PTC Therapeutics (PTC)-sponsored clinical study will continue to receive the same dose/formulation of vatiquinone (unless there has been a change in age and/or weight that meets the criteria for a different dose/formulation as described below; dose/formulation will also be changed if participants meet the criteria for a different dose/formulation during study treatment): If <7 years of age, participants will receive an oral solution (100 milligrams [mg]/milliliter [mL]) 3 times a day (TID) at one of the following doses: 15 mg/kilogram (kg) if body weight <13 kg, or 200 mg if body weight ≥13 kg. If ≥7 years of age, participants will receive a capsule formulation (200 mg) orally TID at one of the following doses: 200 mg if body weight ˂25 kg, or 400 mg if body weight ≥25 kg.
  Interventions: Drug: Vatiquinone

INTERVENTIONS:
Drug: Vatiquinone — Vatiquinone will be administered per dose and schedule specified in the arm.

SUMMARY:
The primary objective of this study is to assess the long-term safety of vatiquinone in participants with Friedreich ataxia (FA) previously exposed to vatiquinone.

DETAILED DESCRIPTION:
This long-term, open-label study will serve as a continued access study for participants with FA who have previously participated in a vatiquinone study. The purpose of this study is to assess continued safety and efficacy of vatiquinone dosing in previously treated participants. This study addresses the medical need for participants to continue vatiquinone with a planned study duration of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants with FA who completed and directly rolled over from a previous vatiquinone clinical study.
* Males and females of childbearing potential must be willing to use an effective method of contraception (for example, implants, injectables, transdermal patches, combined oral contraceptives, barrier methods, and intrauterine devices) from the time consent is signed until 30 days after the last dose of study drug or Early Termination Visit.

Exclusion Criteria:

* Current participation in any other interventional study
* Pregnancy or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Baseline up to 3 years

SECONDARY OUTCOMES:
Change From Baseline in the Modified Friedreich Ataxia Rating Scale (mFARS) and its 4 Subscales (Upright Stability, Upper Limb, Lower Limb, Bulbar) Scores at Year 3 | Baseline, Year 3

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- University of Campinas (UNICAMP) - School of Medical Sciences, Dept of Neurology, São Paulo, Brazil
- Canada (2):
  - Centre de Recherche du Centre Hospitalier de l'Université de Montreal (CRCHUM), Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
- Hôpital Pitié-Salpêtrière, Institut du Cerveau (Paris Brain Institute), Paris, France
- Department of Neurology and Hertie-Institute for Clinical Brain Research German Center of Neurodegenerative Diseases (DZNE), Tübingen, Germany
- Ospedale Pediatrico Bambino Gesu' IRCCS, Roma, Italy
- CBR Neurogenetic Research Clinic, University of Auckland, Auckland, New Zealand
- Hospital Sant Joan de Déu Barcelona Unidad de Enfermedades Neuromusculares, Barcelona, Spain